CLINICAL TRIAL: NCT00006341
Title: Efficacy of Implant-Supported Maxillofacial Prostheses
Brief Title: Dentures and Dental Implants in Treating Patients Undergoing Surgery for Mouth Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000066588; UCLA-HSPC-940205413; UCLA-DEN-1R01DE11255; UCLA-HSPC-940205411; NCI-V00-1606
Record Dates: First submitted 2000-10-04; First posted 2003-05-29 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Head and Neck Cancer
Keywords: stage I lip and oral cavity cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implant (Experimental): A total of 62 patients with early oral cancer will be recruited; in addition, 22 patients requiring a partial maxillectomy and 40 requiring a partial lateral mandibulectomy will be enrolled. The mandibular defects will be reconstructed with fibula free flap surgery. Following a healing period, implants will be placed and permitted to heal unloaded for six months. Conventional dental prostheses will be fabricated and used by patients for at least 16 weeks during Phase I healing before the implants are exposed and loaded. A few weeks after Phase II surgery, the patients will receive implant-supported dental prostheses.
  Interventions: Other: Implant

INTERVENTIONS:
Other: Implant — A total of 62 patients with early oral cancer will be recruited; in addition, 22 patients requiring a partial maxillectomy and 40 requiring a partial lateral mandibulectomy will be enrolled. The mandibular defects will be reconstructed with fibula free flap surgery. Following a healing period, implants will be placed and permitted to heal unloaded for six months. Conventional dental prostheses will be fabricated and used by patients for at least 16 weeks during Phase I healing before the implants are exposed and loaded. A few weeks after Phase II surgery, the patients will receive implant-supported dental prostheses.

SUMMARY:
RATIONALE: The use of dentures and dental implants may help maintain chewing and speaking ability following surgery to remove tumors in the mouth.

PURPOSE: Phase II trial to study the effectiveness of dentures and dental implants in maintaining the ability to chew and speak in patients undergoing surgery for mouth cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether conventional or implant supported dental prostheses and current surgical reconstructive procedures restore oral function and quality of life to pre-cancer surgery levels in patients with early oral cancer.

OUTLINE: Patients complete a series of objective and subjective functional tests, questionnaires, and baseline examinations. Within 1-5 days, patients undergo the composite resection, including reconstructive surgery for the mandibulectomy group. Patients in the maxillectomy group receive an immediate maxillary surgical obturator. Approximately 6 weeks after ablative surgery, some patients receive radiotherapy for 5-7 weeks.

Patients receive 2-4 implants at 12-16 weeks after completion of radiotherapy or 8-16 weeks after ablative surgery. Patients then receive conventional dentures at 4-22 weeks after implant surgery. Implants are exposed during 27-48 weeks after placement and abutments connected for fabricating dental prostheses. Approximately 8 weeks are needed to fabricate the implant supported prosthesis.

Patients complete quality of life and other questionnaires prior to and at 8-21 weeks after surgery, 16 weeks after conventional denture insertion, and then 16 weeks after implant supported prosthesis insertion.

Patients are followed every 6 months for at least 3 years.

PROJECTED ACCRUAL: A total of 62 patients (22 requiring maxillectomy and 40 requiring mandibulectomy) will be accrued for this study within 42 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of early oral cancer lesions requiring one of the following:

  * Partial or total unilateral maxillectomy OR
  * Partial lateral mandibulectomy with or without partial glossectomy
* Edentulous or edentulous in the maxillary arch prior to or after ablative surgery (maxillectomy group)
* Partial mandibulectomy leaving the condyles intact bilaterally (mandibulectomy group)
* Must have sufficient bone in the selected implant sites to accommodate 2-4 implants of at least 10 mm in length
* No temporomandibular dysfunction and/or functionally restrictive opening
* No requirement for total glossectomy, reconstructive maxillary surgery, or maxillary sinus lift
* No requirement for radiotherapy after mandibular reconstructive surgery

PATIENT CHARACTERISTICS:

Age:

* 35 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No oral discomfort that would preclude study
* No complications after ablative or reconstructive surgery that would preclude dental rehabilitation with implants

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior or concurrent radiotherapy of greater than 5,500 cGY to potential implant site

Surgery:

* See Disease Characteristics

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1997-06; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal R. Garrett, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No